CLINICAL TRIAL: NCT01955473
Title: A Japanese Phase I Open-label Dose-escalation Trial of Sym004 Administered as Monotherapy in Japanese Subjects With Advanced Solid Tumors
Brief Title: Japanese Phase 1 Trial of Sym004 in Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EMR 200637-001
Record Dates: First submitted 2013-09-27; First posted 2013-10-07 (Estimated); Results first posted 2017-03-07 (Actual); Last update posted 2017-08-23 (Actual); Status verified 2017-07

CONDITIONS: Solid Tumors
Keywords: Solid tumors; Sym004; Phase 1
MeSH Terms: interventions — futuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sym004 (Experimental)
  Interventions: Drug: Sym004

INTERVENTIONS:
Drug: Sym004 — Part-A (dose-escalation): Sym004 will be administered intravenously either weekly at 6 to 12 milligram per kilogram (mg/kg) or biweekly at 18 mg/kg from Week 1 until unacceptable toxicity, disease progression, or consent withdrawal. Part-B (dose-expansion): After the maximum tolerated dose (MTD) is determined in Part-A, up to 30 additional subjects will continue to receive treatment in Part-B.

SUMMARY:
This trial is to assess the safety and tolerability of Sym004, administered weekly or biweekly as monotherapy in Japanese subjects with advanced solid tumors.This study consisted of two parts, a dose-escalation part ("Part-A") and a dose-expansion part ("Part-B"). In Part-A, Sym004 will be administered weekly or biweekly as monotherapy in Japanese subjects with advanced solid tumors. In Part-B, Sym004 will be administered weekly as monotherapy to Japanese subjects with advanced esophageal squamous cell carcinoma (ESCC) as dose-expansion. A subject will receive Sym004 administration weekly at a dose that will determined to be the MTD or a dose that will lower than the MTD and determined to be appropriate with recommendation by Safety monitoring committee (SMC). The dose going to used in Part-B will be determined after safety confirmation of weekly regimens in Part-A of this trial.

ELIGIBILITY:
Inclusion Criteria:

* Japanese male or female subjects aged greater than or equal to 20 years at the time of informed consent signature
* Histologically or cytologically confirmed cancer
* Refractory or recurrent advanced late stage solid tumors without available therapeutic options which are likely to provide patient benefit (failure and/or intolerance to standard anti-cancer therapy)
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Life expectancy of at least 3 months
* Written informed consent given before any trial-related activities are carried out
* Other protocol defined inclusion criteria could apply

Exclusion Criteria:

* Subjects with symptomatic brain metastases
* Subjects who received total resection or irradiation of the target lesion
* Received any of the following medications within 4 weeks before the first administration of Sym004 at Week 1: cytotoxic or cytostatic anti-cancer therapy, antibody therapy, tyrosine kinase inhibitors, and any investigational agent
* Received vaccine therapy as anticancer treatment within 12 weeks before the first administration of Sym004 at Week 1
* Diarrhea of greater than Grade 1 according to National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 4.03 (v4.03)
* Skin manifestation of greater than Grade 1 according to NCI-CTCAE (v4.03)
* Magnesium of less than 0.9 milligram per deciliter (mg/dL)
* Abnormal organ or bone marrow function as defined in the protocol
* Received immunosuppressive agents (including systemic corticosteroids used at doses above 20 milligram per day (mg/day) of prednisolone or equivalent) within 4 weeks before the first administration of Sym004 at Week 1
* Active severe infection, any other concurrent disease or medical conditions that are deemed to interfere with the conduct of the trial as judged by the Investigator
* Known human immunodeficiency virus (HIV) positive, active Hepatitis B or C, or uncontrolled allergic conditions or allergy to Sym004 or its components
* Clinically significant cardiac disease or concurrent, uncontrolled medical condition
* Known previous Grade 3 to 4 infusion-related reactions, according to NCI-CTCAE (v4.03), with chimeric monoclonal antibodies
* Other protocol defined exclusion criteria could apply

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2013-10-31 (Actual); Primary Completion 2015-10-31 (Actual); Study Completion 2015-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck Serono Co., Ltd. Japan, an business of Merck KGaA, Darmstadt, Germany
Locations (1):
- Please contact the Merck KGaA Communication Center located in, Darmstadt, Germany

REFERENCES:
- [Derived] Kojima T, Yamazaki K, Kato K, Muro K, Hara H, Chin K, Goddemeier T, Kuffel S, Watanabe M, Doi T. Phase I dose-escalation trial of Sym004, an anti-EGFR antibody mixture, in Japanese patients with advanced solid tumors. Cancer Sci. 2018 Oct;109(10):3253-3262. doi: 10.1111/cas.13767. Epub 2018 Sep 25. PMID 30099818

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First/Last subject (informed consent): 30 October 2013/10 Jun 2015. Study completion date: 30 October 2015. Clinical data cut-off: 30 October 2015. The study was conducted by 6 Investigators in 6 sites in Japan.
Pre-assignment Details: A total of 60 subjects were screened for eligibility, out of which and 51 subjects were randomized into the study.
Groups:
- Part A: Sym004 6 mg/kg: Sym004 was administered at a dose of 6 milligram per kilogram (mg/kg) by intravenous infusion weekly until unacceptable toxicity, disease progression, or consent withdrawal, or until the subject met any of the criteria for treatment or trial discontinuation.
- Part A: Sym004 9/6 mg/kg: Sym004 was administered at a dose of 9 mg/kg by intravenous infusion at Week 1 followed by a maintenance dose of 6 mg/kg weekly until unacceptable toxicity, disease progression, or consent withdrawal, or until the subject met any of the criteria for treatment or trial discontinuation.
- Part A: Sym004 12 mg/kg; Part B: Sym004 12 mg/kg: Sym004 was administered at a dose of 12 mg/kg by intravenous infusion weekly until unacceptable toxicity, disease progression, or consent withdrawal, or until the subject met any of the criteria for treatment or trial discontinuation.
- Part A: Sym004 18 mg/kg: Sym004 was administered at a dose of 18 mg/kg by intravenous infusion biweekly until unacceptable toxicity, disease progression, or consent withdrawal, or until the subject met any of the criteria for treatment or trial discontinuation.
Period: Overall Study
Arm/Group | Part A: Sym004 6 mg/kg | Part A: Sym004 9/6 mg/kg | Part A: Sym004 12 mg/kg | Part A: Sym004 18 mg/kg | Part B: Sym004 12 mg/kg
Started | 3 | 6 | 6 | 6 | 30
Completed | 3 | 6 | 6 | 6 | 30
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis set consisted of all subjects (from Parts A and B) who received at least 1 administration of Sym004.
Groups:
- Total: Total of all reporting groups
Arm/Group | Part A: Sym004 6 mg/kg | Part A: Sym004 9/6 mg/kg | Part A: Sym004 12 mg/kg | Part A: Sym004 18 mg/kg | Part B: Sym004 12 mg/kg | Total
Number analyzed (Participants) | 3 | 6 | 6 | 6 | 30 | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.7 (3.51) | 62.5 (5.09) | 66.5 (5.96) | 59.0 (9.32) | 61.2 (7.20) | 61.6 (7.03)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3 | 0 | 6 | 12
  Male | 1 | 5 | 3 | 6 | 24 | 39

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Dose Limiting Toxicities (DLTs) Determined in Part-A
Description: DLT: any of the following National Cancer Institute Common Toxicity Criteria for Adverse Events (NCI-CTCAE) Grade 4 hematologic or Grade 3/4 non-hematologic toxicities that occurred during DLT observation period of Part A, and were considered by Investigator to be at least possibly related to study treatment, and confirmed by Safety Monitoring Committee. Hematological toxicities: Grade 4 neutropenia, febrile neutropenia, Grade 4 thrombocytopenia, Grade 3 thrombocytopenia with bleeding episodes. Nonhematological toxicities: Grade 3 or higher non-hematological toxicity with exception of Grade 3 fatigue/skin toxicity; Grade 3 nausea/vomiting without appropriate prophylactic therapy; Grade 3 diarrhoea recovered within 2 days with adequate treatment or did not accompany fever/dehydration; Grade 3 or 4 laboratory liver parameter abnormalities with duration of less than 3 days.
Time Frame: Week 1 up to Week 4 (Part A)
Population: DLT Analysis Set consisted of all subjects who received at least 3 of 4 weekly administrations (for weekly dosing cohort) or who received 2 biweekly administrations (for biweekly dosing cohort) and experienced a DLT during DLT observation period.
Measure: Number; unit: subjects
Arm/Group | Part A: Sym004 6 mg/kg | Part A: Sym004 9/6 mg/kg | Part A: Sym004 12 mg/kg | Part A: Sym004 18 mg/kg
Number analyzed (Participants) | 3 | 6 | 6 | 6
subjects | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Subjects With Treatment-emergent Adverse (TEAEs), Serious TEAEs, TEAEs Leading to Discontinuation or TEAEs Leading to Death
Description: An adverse event (AE) was defined as any untoward medical occurrence in a subject which does not necessarily have a causal relationship with the treatment. An AE was any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with use of a medicinal product, whether or not considered related to the medicinal product. A serious adverse event (SAE) was an AE that resulted in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial or prolonged inpatient hospitalization; congenital anomaly/birth defect or was otherwise considered medically important. AEs were considered treatment emergent if they started on or after the day of first administration of the Sym004 or if they started prior to administration but worsened after receiving the first dose of treatment.
Time Frame: Baseline up to 4 weeks after the last Sym004 administration, up to a maximum of 41.1 weeks
Population: Safety analysis set consisted of all subjects (from Parts A and B) who received at least 1 administration of Sym004.
Measure: Number; unit: subjects
Arm/Group | Part A: Sym004 6 mg/kg | Part A: Sym004 9/6 mg/kg | Part A: Sym004 12 mg/kg | Part A: Sym004 18 mg/kg | Part B: Sym004 12 mg/kg
Number analyzed (Participants) | 3 | 6 | 6 | 6 | 30
subjects
  TEAEs | 3 | 6 | 6 | 6 | 30
  Serious TEAEs | 0 | 0 | 2 | 0 | 9
  TEAE leading to Discontinuation | 0 | 0 | 0 | 0 | 4
  TEAEs Leading to Death | 0 | 0 | 0 | 0 | 3

3. Secondary Outcome: Area Under Concentration-time Curve (AUC) From Start of First Infusion to 168 Hours (AUC0-168h) at Week 1: Single Dose
Description: Sym004 is a mixture of two mouse-human chimeric immunoglobulin G1 anti-epidermal growth factor receptor (EGFR) monoclonal antibodies (called monoclonal antibodies [mAb] 992 and mAb 1024). Here AUC are presented for both monoclonal antibodies.
Time Frame: Pre-infusion, end of infusion, 4, 8, 12, 24, 48 and 168 hours post-infusion at Week 1
Population: The Pharmacokinetics (PK) Analysis Set consisted of all subjects (from Parts A and B) who received at least 1 administration of Sym004 and who provided sufficient data for a concentration time profile for Sym004. Here "Number of Participants Analyzed" signifies those subjects who were evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg*h/mL
Arm/Group | Part A: Sym004 6 mg/kg | Part A: Sym004 9/6 mg/kg | Part A: Sym004 12 mg/kg | Part A: Sym004 18 mg/kg | Part B: Sym004 12 mg/kg
Number analyzed (Participants) | 3 | 6 | 6 | 6 | 7
μg*h/mL
  mAb992 | 3685.5 (38.1) | 5893.1 (33.3) | 8957.3 (29.3) | 12783 (26.0) | 7073.5 (15.1)
  mAb1024 | 4109.0 (25.6) | 6572.1 (30.5) | 10213 (24.1) | 15917 (30.6) | 10336 (27.4)

4. Secondary Outcome: Area Under Concentration-time Curve (AUC) From Start of First Infusion to 168 Hours (AUC0-168h) for the Weekly Regimen at Week 4: Multiple Dose
Description: Sym004 is a mixture of two mouse-human chimeric immunoglobulin G1 anti-epidermal growth factor receptor (EGFR) monoclonal antibodies (called monoclonal antibodies [mAb] 992 and mAb 1024). Here AUC are presented for both monoclonal antibodies. Results were to be assessed for weekly dosing cohorts (Part A: Sym004 6 mg/kg, Part A: Sym004 9/6 mg/kg, Part A: Sym004 12 mg/kg, Part B: Sym004 12 mg/kg) only.
Time Frame: Pre-infusion, end of infusion, 4, 8, 12, 24, and 168 hours post-infusion at Week 4
Population: The PK Analysis Set consisted of all subjects (from Parts A and B) who received at least 1 administration of Sym004 and who provided sufficient data for a concentration time profile for Sym004. Here "Number of Participants Analyzed" =subjects who were evaluable for this outcome and "n" =subjects who were evaluable for specified monoclonal antibody.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg*h/mL
Arm/Group | Part A: Sym004 6 mg/kg | Part A: Sym004 9/6 mg/kg | Part A: Sym004 12 mg/kg | Part B: Sym004 12 mg/kg
Number analyzed (Participants) | 2 | 5 | 6 | 5
μg*h/mL
  mAb992 (n=2, 5, 6, 5) | NA (NA) — Geometric mean and Geometric coefficient of variation was not estimable if evaluable subjects were less than 3 as per the planned decision because only 2 collected values were not sufficient to calculate a reliable estimation | 7111.1 (41.7) | 15298 (41.4) | 13053 (18.7)
  mAb1024 (n=2, 4, 6, 5) | NA (NA) — Geometric mean and Geometric coefficient of variation was not estimable if evaluable subjects were less than 3 as per the planned decision because only 2 collected values were not sufficient to calculate a reliable estimation | 9738.5 (36.8) | 21422 (45.5) | 22016 (32.2)

5. Secondary Outcome: Dose Normalized Area Under Concentration-time Curve (AUC) From Start of First Infusion to 168 Hours (AUC0-168h) at Week 1: Single Dose
Description: Sym004 is a mixture of two mouse-human chimeric immunoglobulin G1 anti-epidermal growth factor receptor (EGFR) monoclonal antibodies (called monoclonal antibodies [mAb] 992 and mAb 1024). Here dose normalized AUC are presented for both monoclonal antibodies. Dose normalized AUC for AUC0-168 was calculated as AUC(0-168)/Dose.
Time Frame: Pre-infusion, end of infusion, 4, 8, 12, 24, 48 and 168 hours post-infusion at Week 1
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg*h/mL/mg
Arm/Group | Part A: Sym004 6 mg/kg | Part A: Sym004 9/6 mg/kg | Part A: Sym004 12 mg/kg | Part A: Sym004 18 mg/kg | Part B: Sym004 12 mg/kg
Number analyzed (Participants) | 3 | 6 | 6 | 6 | 7
μg*h/mL/mg
  mAb992 | 22.50 (29.5) | 23.24 (30.7) | 25.79 (18.0) | 21.69 (24.8) | 22.70 (17.5)
  mAb1024 | 25.09 (20.1) | 25.91 (27.7) | 29.41 (11.1) | 27.01 (26.0) | 33.17 (27.8)

6. Secondary Outcome: Dose Nornamized Area Under Concentration-time Curve (AUC) From Start of First Infusion to 168 Hours (AUC0-168h) for the Weekly Regimen at Week 4: Multiple Dose
Description: Sym004 is a mixture of two mouse-human chimeric immunoglobulin G1 anti-epidermal growth factor receptor (EGFR) monoclonal antibodies (called monoclonal antibodies [mAb] 992 and mAb 1024). Here dose normalized AUC are presented for both monoclonal antibodies. Dose normalized AUC for AUC0-168 was calculated as AUC(0-168)/Dose. Results were to be assessed for weekly dosing cohorts (Part A: Sym004 6 mg/kg, Part A: Sym004 9/6 mg/kg, Part A: Sym004 12 mg/kg, Part B: Sym004 12 mg/kg) only.
Time Frame: Pre-infusion, end of infusion, 4, 8, 12, 24, and 168 hours post-infusion at Week 4
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg*h/mL/mg
Arm/Group | Part A: Sym004 6 mg/kg | Part A: Sym004 9/6 mg/kg | Part A: Sym004 12 mg/kg | Part B: Sym004 12 mg/kg
Number analyzed (Participants) | 2 | 5 | 6 | 5
μg*h/mL/mg
  mAb992 (n= 2, 5, 6, 5) | NA (NA) — Geometric mean and Geometric coefficient of variation was not estimable if evaluable subjects were less than 3 as per the planned decision because only 2 collected values were not sufficient to calculate a reliable estimation | 43.90 (27.3) | 43.45 (29.3) | 42.38 (15.0)
  mAb1024 (n= 2, 4, 6, 5) | NA (NA) — Geometric mean and Geometric coefficient of variation was not estimable if evaluable subjects were less than 3 as per the planned decision because only 2 collected values were not sufficient to calculate a reliable estimation | 59.12 (30.6) | 60.85 (32.9) | 72.36 (28.2)

7. Secondary Outcome: Area Under Concentration-time Curve (AUC) From Start of First Infusion to 336 Hours (AUC0-336hours) For the Biweekly Regimen at Week 1: Single Dose
Description: Sym004 is a mixture of two mouse-human chimeric immunoglobulin G1 anti-epidermal growth factor receptor (EGFR) monoclonal antibodies (called monoclonal antibodies [mAb] 992 and mAb 1024). Here AUC are presented for both monoclonal antibodies. Results were to be assessed for biweekly dosing cohort (Part A: Sym004 18 mg/kg) only.
Time Frame: Pre-infusion, end of infusion, 4, 8, 12, 24, 48, 168, 336 hours post-infusion at Week 1
Population: The PK Analysis Set consisted of all subjects who received at least 1 administration of Sym004 and who provided sufficient data for a concentration time profile for Sym004.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg*h/mL
Arm/Group | Part A: Sym004 18 mg/kg
Number analyzed (Participants) | 6
μg*h/mL
  mAb992 | 17318 (27.0)
  mAb1024 | 22458 (29.7)

8. Secondary Outcome: Area Under Concentration-time Curve (AUC) From Start of First Infusion to 336 Hours (AUC0-336hours) For the Biweekly Regimen at Week 5: Multiple Dose
Description: as for outcome 7
Time Frame: Pre-infusion, end of infusion, 4, 8, 12, 24, 168 and 336 hours post-infusion at Week 5
Population: The PK Analysis Set consisted of all subjects who received at least 1 administration of Sym004 and who provided sufficient data for a concentration time profile for Sym004. Here, "Number of Participants Analyzed" signifies those subjects who were evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg*h/mL
Arm/Group | Part A: Sym004 18 mg/kg
Number analyzed (Participants) | 5
μg*h/mL
  mAb992 | 24755 (31.8)
  mAb1024 | 32336 (30.8)

9. Secondary Outcome: Dose Normalized Area Under Concentration-time Curve (AUC) From Start of First Infusion to 336 Hours (AUC0-336hours) For the Biweekly Regimen at Week 1: Single Dose
Description: Sym004 is a mixture of two mouse-human chimeric immunoglobulin G1 anti-epidermal growth factor receptor (EGFR) monoclonal antibodies (called monoclonal antibodies [mAb] 992 and mAb 1024). Here dose normalized AUC are presented for both monoclonal antibodies. Results were to be assessed for biweekly dosing cohort (Part A: Sym004 18 mg/kg) only. Dose normalized AUC for AUC0-336 was calculated as AUC(0-336)/Dose.
Time Frame: Pre-infusion, end of infusion, 4, 8, 12, 24, 48, 168, 336 hours post-infusion at Week 1
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg*h/mL/mg
Arm/Group | Part A: Sym004 18 mg/kg
Number analyzed (Participants) | 6
μg*h/mL/mg
  mAb992 | 29.39 (27.1)
  mAb1024 | 38.11 (26.9)

10. Secondary Outcome: Dose Normalized Area Under Concentration-time Curve (AUC) From Start of First Infusion to 336 Hours (AUC0-336hours) For the Biweekly Regimen at Week 5: Multiple Dose
Description: as for outcome 9
Time Frame: Pre-infusion, end of infusion, 4, 8, 12, 24, 168 and 336 hours post-infusion at Week 5
Population: as for outcome 8
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg*h/mL/mg
Arm/Group | Part A: Sym004 18 mg/kg
Number analyzed (Participants) | 5
μg*h/mL/mg
  mAb992 | 42.45 (29.9)
  mAb1024 | 55.46 (25.7)

11. Secondary Outcome: Area Under Concentration-time Curve (AUC) From Start of First Infusion to Infinity (AUC0-inf) For the Biweekly Regimen at Week 1: Single Dose
Description: as for outcome 7
Time Frame: Pre-infusion, end of infusion, 4, 8, 12, 24, and 48 hours post-infusion at Week 1
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg*h/mL
Arm/Group | Part A: Sym004 18 mg/kg
Number analyzed (Participants) | 6
μg*h/mL
  mAb992 | 19896 (28.9)
  mAb1024 | 27554 (30.7)

12. Secondary Outcome: Area Under Concentration-time Curve (AUC) From Start of First Infusion to Infinity (AUC0-inf) For the Biweekly Regimen at Week 5: Multiple Dose
Description: as for outcome 7
Time Frame: Pre-infusion, end of infusion, 4, 8, 12 and 24 hours post-infusion at Week 5
Population: as for outcome 8
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg*h/mL
Arm/Group | Part A: Sym004 18 mg/kg
Number analyzed (Participants) | 5
μg*h/mL
  mAb992 | 30127 (36.6)
  mAb1024 | 43308 (37.8)

13. Secondary Outcome: Dose Normalized Area Under Concentration-time Curve (AUC) From Start of First Infusion to Infinity (AUC0-inf) at Week 1: Single Dose
Description: Sym004 is a mixture of two mouse-human chimeric immunoglobulin G1 anti-epidermal growth factor receptor (EGFR) monoclonal antibodies (called monoclonal antibodies [mAb] 992 and mAb 1024). Here dose normalized AUC are presented for both monoclonal antibodies. Dose normalized AUC for AUC0-inf was calculated as AUC(0-inf)/Dose.
Time Frame: Pre-infusion, end of infusion, 4, 8, 12, 24, and 48 hours post-infusion at Week 1
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg*h/mL/mg
Arm/Group | Part A: Sym004 6 mg/kg | Part A: Sym004 9/6 mg/kg | Part A: Sym004 12 mg/kg | Part A: Sym004 18 mg/kg | Part B: Sym004 12 mg/kg
Number analyzed (Participants) | 3 | 6 | 6 | 6 | 7
μg*h/mL/mg
  mAb992 (3, 6, 6, 6, 7) | 27.30 (26.7) | 30.33 (37.7) | 34.471 (22.5) | 33.77 (30.3) | 31.05 (24.6)
  mAb1024 (3, 6, 6, 6, 6) | 31.86 (21.9) | 36.20 (37.4) | 43.41 (23.1) | 46.77 (30.9) | 47.48 (17.5)

14. Secondary Outcome: Dose Normalized Area Under Concentration-time Curve (AUC) From Start of First Infusion to Infinity (AUC0-inf) for the Weekly Regimen at Week 4: Multiple Dose
Description: Sym004 is a mixture of two mouse-human chimeric immunoglobulin G1 anti-epidermal growth factor receptor (EGFR) monoclonal antibodies (called monoclonal antibodies [mAb] 992 and mAb 1024). Here dose normalized AUC are presented for both monoclonal antibodies. Weekly dosing cohorts (Part A: Sym004 6 mg/kg, Part A: Sym004 9/6 mg/kg, Part A: Sym004 12 mg/kg, Part B: Sym004 12 mg/kg) were only applicable for Week 4 assessment. Biweekly dosing cohort (Part A: Sym004 18 mg/kg) was not applicable for Week 4 assessment. Dose normalized AUC for AUC0-inf was calculated as AUC(0-inf)/Dose.
Time Frame: Pre-infusion, end of infusion, 4, 8, 12, 24 hours post-infusion at Week 4
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg*h/mL/mg
Arm/Group | Part A: Sym004 6 mg/kg | Part A: Sym004 9/6 mg/kg | Part A: Sym004 12 mg/kg | Part B: Sym004 12 mg/kg
Number analyzed (Participants) | 2 | 5 | 6 | 5
μg*h/mL/mg
  mAb992 (n= 1, 5, 6, 5) | NA (NA) — Geometric mean and Geometric coefficient of variation was not estimable if evaluable subjects were less than 3 as per the planned decision because only 2 collected values were not sufficient to calculate a reliable estimation | 59.65 (37.3) | 77.86 (65.2) | 72.22 (17.1)
  mAb1024 (n= 2, 4, 6, 4) | NA (NA) — Geometric mean and Geometric coefficient of variation was not estimable if evaluable subjects were less than 3 as per the planned decision because only 2 collected values were not sufficient to calculate a reliable estimation | 94.91 (44.7) | 118.1 (57.5) | 136.9 (46.8)

15. Secondary Outcome: Dose Normalized Area Under Concentration-time Curve (AUC) From Start of First Infusion to Infinity (AUC0-inf) For the Biweekly Regimen at Week 5: Multiple Dose
Description: Sym004 is a mixture of two mouse-human chimeric immunoglobulin G1 anti-epidermal growth factor receptor (EGFR) monoclonal antibodies (called monoclonal antibodies [mAb] 992 and mAb 1024). Here dose normalized AUC are presented for both monoclonal antibodies. Weekly dosing cohorts (Part A: Sym004 6 mg/kg, Part A: Sym004 9/6 mg/kg, Part A: Sym004 12 mg/kg, Part B: Sym004 12 mg/kg) were not applicable for Week 5 assessment. Biweekly dosing cohort (Part A: Sym004 18 mg/kg) was only applicable for Week 5 assessment. Dose normalized AUC for AUC0-inf was calculated as AUC(0-inf)/Dose.
Time Frame: Pre-infusion, end of infusion, 4, 8, 12, 24 hours post-infusion at Week 5
Population: The PK Analysis Set consisted of all subjects who received at least 1 administration of Sym004 and who provided sufficient data for a concentration time profile for Sym004. Here "Number of Participants Analyzed" signifies those subjects who were evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg*h/mL/mg
Arm/Group | Part A: Sym004 18 mg/kg
Number analyzed (Participants) | 5
μg*h/mL/mg
  mAb992 | 51.67 (36.2)
  mAb1024 | 74.28 (36.3)

16. Secondary Outcome: Terminal Half-life (t1/2) of Sym004 at Week 1: Single Dose
Description: Terminal half-life was defined as the time required for the serum concentration of drug to decrease 50 percent in the final stage of its elimination. Sym004 is a mixture of two mouse-human chimeric immunoglobulin G1 anti-epidermal growth factor receptor (EGFR) monoclonal antibodies (called monoclonal antibodies [mAb] 992 and mAb 1024). Terminal t1/2 are presented for both monoclonal antibodies.
Time Frame: Pre-infusion, end of infusion, 4, 8, 12, 24, 48 hours post-infusion at Week 1
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Part A: Sym004 6 mg/kg | Part A: Sym004 9/6 mg/kg | Part A: Sym004 12 mg/kg | Part A: Sym004 18 mg/kg | Part B: Sym004 12 mg/kg
Number analyzed (Participants) | 3 | 6 | 6 | 6 | 7
hours
  mAb992 (n= 3,6,6,6,7) | 66.478 (10.0) | 79.041 (18.8) | 82.865 (21.1) | 111.69 (18.9) | 87.257 (21.1)
  mAb1024 (n= 3,6,6,6,6) | 74.075 (8.8) | 91.303 (21.7) | 100.05 (24.3) | 134.48 (27.8) | 100.57 (34.8)

17. Secondary Outcome: Terminal Half-life (t1/2) of Sym004 for the Weekly Regimen at Week 4: Multiple Dose
Description: Terminal half-life was defined as the time required for the serum concentration of drug to decrease 50 percent in the final stage of its elimination. Sym004 is a mixture of two mouse-human chimeric immunoglobulin G1 anti-epidermal growth factor receptor (EGFR) monoclonal antibodies (called monoclonal antibodies [mAb] 992 and mAb 1024). Terminal t1/2 are presented for both monoclonal antibodies. Weekly dosing cohorts (Part A: Sym004 6 mg/kg, Part A: Sym004 9/6 mg/kg, Part A: Sym004 12 mg/kg, Part B: Sym004 12 mg/kg) were only applicable for Week 4 assessment. Biweekly dosing cohort (Part A: Sym004 18 mg/kg) was not applicable for Week 4 assessment.
Time Frame: Pre-infusion, end of infusion, 4, 8, 12, 24 hours post-infusion at Week 4
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Part A: Sym004 6 mg/kg | Part A: Sym004 9/6 mg/kg | Part A: Sym004 12 mg/kg | Part B: Sym004 12 mg/kg
Number analyzed (Participants) | 2 | 5 | 6 | 5
hours
  mAb992 (n= 1, 5, 6, 5) | NA (NA) — Geometric mean and Geometric coefficient of variation was not estimable if evaluable subjects were less than 3 as per the planned decision because only 2 collected values were not sufficient to calculate a reliable estimation | 85.228 (24.4) | 135.98 (52.5) | 132.14 (13.9)
  mAb1024 (n= 2, 4, 6, 4) | NA (NA) — Geometric mean and Geometric coefficient of variation was not estimable if evaluable subjects were less than 3 as per the planned decision because only 2 collected values were not sufficient to calculate a reliable estimation | 117.8 (27.5) | 155.9 (37.4) | 163.8 (27.5)

18. Secondary Outcome: Terminal Half-life (t1/2) of Sym004 For the Biweekly Regimen at Week 5: Multiple Dose
Description: Terminal half-life was defined as the time required for the serum concentration of drug to decrease 50 percent in the final stage of its elimination. Sym004 is a mixture of two mouse-human chimeric immunoglobulin G1 anti-epidermal growth factor receptor (EGFR) monoclonal antibodies (called monoclonal antibodies [mAb] 992 and mAb 1024). Terminal t1/2 are presented for both monoclonal antibodies. Weekly dosing cohorts (Part A: Sym004 6 mg/kg, Part A: Sym004 9/6 mg/kg, Part A: Sym004 12 mg/kg, Part B: Sym004 12 mg/kg) were not applicable for Week 5 assessment. Biweekly dosing cohort (Part A: Sym004 18 mg/kg) was only applicable for Week 5 assessment.
Time Frame: Pre-infusion, end of infusion, 4, 8, 12, 24 hours post-infusion at Week 5
Population: as for outcome 15
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Part A: Sym004 18 mg/kg
Number analyzed (Participants) | 5
hours
  mAb992 | 130.39 (26.4)
  mAb1024 | 163.6 (36.3)

19. Secondary Outcome: Clearance (CL) of Sym004 at Week 1: Single Dose
Description: Clearance of a drug was a measure of the rate at which a drug was metabolized or eliminated by normal biological processes. Sym004 is a mixture of two mouse-human chimeric immunoglobulin G1 anti-epidermal growth factor receptor (EGFR) monoclonal antibodies (called monoclonal antibodies [mAb] 992 and mAb 1024). CL are presented for both monoclonal antibodies.
Time Frame: Pre-infusion, end of infusion, 4, 8, 12, 24, 48 hours post-infusion at Week 1
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter/hour
Arm/Group | Part A: Sym004 6 mg/kg | Part A: Sym004 9/6 mg/kg | Part A: Sym004 12 mg/kg | Part A: Sym004 18 mg/kg | Part B: Sym004 12 mg/kg
Number analyzed (Participants) | 3 | 6 | 6 | 6 | 7
Liter/hour
  mAb992 (n= 3,6,6,6,7) | 0.036626 (26.7) | 0.032967 (37.7) | 0.029012 (22.5) | 0.029615 (30.3) | 0.032202 (24.6)
  mAb1024 (n= 3,6,6,6,6) | 0.031385 (21.9) | 0.027622 (37.4) | 0.023033 (23.1) | 0.021383 (30.9) | 0.021058 (17.6)

20. Secondary Outcome: Clearance at Steady-state (CLss) of Sym004 for the Weekly Regimen at Week 4: Multiple Dose
Description: Clearance at steady state was reported. Clearance of a drug was a measure of the rate at which a drug was metabolized or eliminated by normal biological processes. Sym004 is a mixture of two mouse-human chimeric immunoglobulin G1 anti-epidermal growth factor receptor (EGFR) monoclonal antibodies (called monoclonal antibodies [mAb] 992 and mAb 1024). CLss are presented for both monoclonal antibodies. Weekly dosing cohorts (Part A: Sym004 6 mg/kg, Part A: Sym004 9/6 mg/kg, Part A: Sym004 12 mg/kg, Part B: Sym004 12 mg/kg) were only applicable for Week 4 assessment. Biweekly dosing cohort (Part A: Sym004 18 mg/kg) was not applicable for Week 4 assessment.
Time Frame: Pre-infusion, end of infusion, 4, 8, 12, 24 hours post-infusion at Week 4
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter/hour
Arm/Group | Part A: Sym004 6 mg/kg | Part A: Sym004 9/6 mg/kg | Part A: Sym004 12 mg/kg | Part B: Sym004 12 mg/kg
Number analyzed (Participants) | 2 | 5 | 6 | 5
Liter/hour
  mAb992 (n= 2, 5, 6, 5) | NA (NA) — Geometric mean and Geometric coefficient of variation was not estimable if evaluable subjects were less than 3 as per the planned decision because only 2 collected values were not sufficient to calculate a reliable estimation | 0.022778 (27.3) | 0.023015 (29.3) | 0.023589 (15.0)
  mAb1024 (n= 2, 4, 6, 4) | NA (NA) — Geometric mean and Geometric coefficient of variation was not estimable if evaluable subjects were less than 3 as per the planned decision because only 2 collected values were not sufficient to calculate a reliable estimation | 0.017 (30.6) | 0.016 (32.9) | 0.014 (28.2)

21. Secondary Outcome: Clearance at Steady-state (CLss) of Sym004 for the Biweekly Regimen at Week 5: Multiple Dose
Description: Clearance at steady state was reported. Clearance of a drug was a measure of the rate at which a drug was metabolized or eliminated by normal biological processes. Sym004 is a mixture of two mouse-human chimeric immunoglobulin G1 anti-epidermal growth factor receptor (EGFR) monoclonal antibodies (called monoclonal antibodies [mAb] 992 and mAb 1024). CLss are presented for both monoclonal antibodies. Weekly dosing cohorts (Part A: Sym004 6 mg/kg, Part A: Sym004 9/6 mg/kg, Part A: Sym004 12 mg/kg, Part B: Sym004 12 mg/kg) were not applicable for Week 5 assessment. Biweekly dosing cohort (Part A: Sym004 18 mg/kg) was only applicable for Week 5 assessment.
Time Frame: Pre-infusion, end of infusion, 4, 8, 12, 24 hours post-infusion at Week 5
Population: as for outcome 15
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter/hour
Arm/Group | Part A: Sym004 18 mg/kg
Number analyzed (Participants) | 5
Liter/hour
  mAb992 | 0.023552 (29.9)
  mAb1024 | 0.018 (25.6)

22. Secondary Outcome: Volume of Distribution at the Elimination Phase (Vz) of Sym004 at Week 1: Single Dose
Description: Volume of distribution was defined as the theoretical volume in which the total amount of drug needed to be uniformly distributed to produce the desired serum concentration of a drug. Sym004 is a mixture of two mouse-human chimeric immunoglobulin G1 anti-epidermal growth factor receptor (EGFR) monoclonal antibodies (called monoclonal antibodies [mAb] 992 and mAb 1024). Vz are presented for both monoclonal antibodies.
Time Frame: Pre-infusion, end of infusion, 4, 8, 12, 24, 48 hours post-infusion at Week 1
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter
Arm/Group | Part A: Sym004 6 mg/kg | Part A: Sym004 9/6 mg/kg | Part A: Sym004 12 mg/kg | Part A: Sym004 18 mg/kg | Part B: Sym004 12 mg/kg
Number analyzed (Participants) | 3 | 6 | 6 | 6 | 7
Liter
  mAb992 (n= 3,6,6,6,7) | 3.5130 (36.1) | 3.7593 (21.9) | 3.4688 (17.8) | 4.7726 (23.3) | 4.0536 (10.8)
  mAb1024 (n= 3,6,6,6,6) | 3.3543 (16.7) | 3.6384 (17.6) | 3.3245 (3.4) | 4.1483 (29.1) | 3.0558 (47.0)

23. Secondary Outcome: Volume of Distribution at Steady State (Vss) of Sym004 for the Weekly Regimen at Week 4: Multiple Dose
Description: Volume of distribution was defined as the theoretical volume in which the total amount of drug needed to be uniformly distributed to produce the desired serum concentration of a drug. Sym004 is a mixture of two mouse-human chimeric immunoglobulin G1 anti-epidermal growth factor receptor (EGFR) monoclonal antibodies (called monoclonal antibodies [mAb] 992 and mAb 1024). Vss are presented for both monoclonal antibodies. Weekly dosing cohorts (Part A: Sym004 6 mg/kg, Part A: Sym004 9/6 mg/kg, Part A: Sym004 12 mg/kg, Part B: Sym004 12 mg/kg) were only applicable for Week 4 assessment. Biweekly dosing cohort (Part A: Sym004 18 mg/kg) was not applicable for Week 4 assessment.
Time Frame: Pre-infusion, end of infusion, 4, 8, 12, 24 hours post-infusion at Week 4
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter
Arm/Group | Part A: Sym004 6 mg/kg | Part A: Sym004 9/6 mg/kg | Part A: Sym004 12 mg/kg | Part B: Sym004 12 mg/kg
Number analyzed (Participants) | 2 | 5 | 6 | 5
Liter
  mAb992 (n= 1, 5, 6, 5) | NA (NA) — Geometric mean and Geometric coefficient of variation was not estimable if evaluable subjects were less than 3 as per the planned decision because only 2 collected values were not sufficient to calculate a reliable estimation | 2.7931 (15.4) | 4.4777 (26.2) | 4.4383 (17.9)
  mAb1024 (n= 2, 4, 6, 4) | NA (NA) — Geometric mean and Geometric coefficient of variation was not estimable if evaluable subjects were less than 3 as per the planned decision because only 2 collected values were not sufficient to calculate a reliable estimation | 2.85 (20.6) | 3.71 (21.3) | 3.40 (24.9)

24. Secondary Outcome: Volume of Distribution at Steady State (Vss) of Sym004 for the Biweekly Regimen at Week 5: Multiple Dose
Description: Volume of distribution was defined as the theoretical volume in which the total amount of drug needed to be uniformly distributed to produce the desired serum concentration of a drug. Sym004 is a mixture of two mouse-human chimeric immunoglobulin G1 anti-epidermal growth factor receptor (EGFR) monoclonal antibodies (called monoclonal antibodies [mAb] 992 and mAb 1024). Vss are presented for both monoclonal antibodies. Weekly dosing cohorts (Part A: Sym004 6 mg/kg, Part A: Sym004 9/6 mg/kg, Part A: Sym004 12 mg/kg, Part B: Sym004 12 mg/kg) were not applicable for Week 5 assessment. Biweekly dosing cohort (Part A: Sym004 18 mg/kg) was only applicable for Week 5 assessment.
Time Frame: Pre-infusion, end of infusion, 4, 8, 12, 24 hours post-infusion at Week 5
Population: as for outcome 15
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter
Arm/Group | Part A: Sym004 18 mg/kg
Number analyzed (Participants) | 5
Liter
  mAb992 | 4.3988 (24.4)
  mAb1024 | 4.20 (27.7)

25. Secondary Outcome: Maximum Serum Concentration (Cmax) of Sym004 at Week 1: Single Dose
Description: Sym004 is a mixture of two mouse-human chimeric immunoglobulin G1 anti-epidermal growth factor receptor (EGFR) monoclonal antibodies (called monoclonal antibodies [mAb] 992 and mAb 1024). Cmax are presented for both monoclonal antibodies.
Time Frame: Pre-infusion, end of infusion, 4, 8, 12, 24, 48 hours post-infusion at Week 1
Population: The PK Analysis Set consisted of all subjects (from Parts A and B) who received at least 1 administration of Sym004 and who provided sufficient data for a concentration time profile for Sym004. Here "Number of Participants Analyzed" signifies those subjects who were evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram per milliliter (μg/mL)
Arm/Group | Part A: Sym004 6 mg/kg | Part A: Sym004 9/6 mg/kg | Part A: Sym004 12 mg/kg | Part A: Sym004 18 mg/kg | Part B: Sym004 12 mg/kg
Number analyzed (Participants) | 3 | 6 | 6 | 6 | 7
microgram per milliliter (μg/mL)
  mAb992 | 50.131 (29.2) | 85.088 (25.3) | 120.37 (33.6) | 157.71 (18.6) | 88.589 (15.0)
  mAb1024 | 54.660 (15.6) | 89.443 (26.2) | 116.18 (31.2) | 187.03 (23.9) | 146.92 (56.3)

26. Secondary Outcome: Maximum Serum Concentration (Cmax) of Sym004 for the Weekly Regimen at Week 4: Multiple Dose
Description: Sym004 is a mixture of two mouse-human chimeric immunoglobulin G1 anti-epidermal growth factor receptor (EGFR) monoclonal antibodies (called monoclonal antibodies [mAb] 992 and mAb 1024). Cmax are presented for both monoclonal antibodies. Weekly dosing cohorts (Part A: Sym004 6 mg/kg, Part A: Sym004 9/6 mg/kg, Part A: Sym004 12 mg/kg, Part B: Sym004 12 mg/kg) were only applicable for Week 4 assessment. Biweekly dosing cohort (Part A: Sym004 18 mg/kg) was not applicable for Week 4 assessment.
Time Frame: Pre-infusion, end of infusion, 4, 8, 12, 24 hours post-infusion at Week 4
Population: as for outcome 25
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Arm/Group | Part A: Sym004 6 mg/kg | Part A: Sym004 9/6 mg/kg | Part A: Sym004 12 mg/kg | Part B: Sym004 12 mg/kg
Number analyzed (Participants) | 3 | 6 | 6 | 6
μg/mL
  mAb992 | 76.094 (16.4) | 86.763 (34.0) | 181.62 (31.6) | 143.79 (23.4)
  mAb1024 | 89.26 (10.2) | 91.70 (33.4) | 221.3 (21.1) | 231.9 (32.8)

27. Secondary Outcome: Maximum Serum Concentration (Cmax) of Sym004 for the Biweekly Regimen at Week 5: Multiple Dose
Description: Sym004 is a mixture of two mouse-human chimeric immunoglobulin G1 anti-epidermal growth factor receptor (EGFR) monoclonal antibodies (called monoclonal antibodies [mAb] 992 and mAb 1024). Cmax are presented for both monoclonal antibodies. Weekly dosing cohorts (Part A: Sym004 6 mg/kg, Part A: Sym004 9/6 mg/kg, Part A: Sym004 12 mg/kg, Part B: Sym004 12 mg/kg) were not applicable for Week 5 assessment. Biweekly dosing cohort (Part A: Sym004 18 mg/kg) was only applicable for Week 5 assessment.
Time Frame: Pre-infusion, end of infusion, 4, 8, 12, 24 hours post-infusion at Week 5
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Arm/Group | Part A: Sym004 18 mg/kg
Number analyzed (Participants) | 6
μg/mL
  mAb992 | 187.40 (24.3)
  mAb1024 | 224.0 (24.7)

28. Secondary Outcome: Dose Normalized Maximum Serum Concentration (Cmax) of Sym004 at Week 1: Single Dose
Description: Sym004 is a mixture of two mouse-human chimeric immunoglobulin G1 anti-epidermal growth factor receptor (EGFR) monoclonal antibodies (called monoclonal antibodies [mAb] 992 and mAb 1024). Dose Normalized Cmax are presented for both monoclonal antibodies. Dose normalized Cmax was calculated as Cmax/Dose.
Time Frame: Pre-infusion, end of infusion, 4, 8, 12, 24, 48 hours post-infusion at Week 1
Population: as for outcome 25
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL/mg
Arm/Group | Part A: Sym004 6 mg/kg | Part A: Sym004 9/6 mg/kg | Part A: Sym004 12 mg/kg | Part A: Sym004 18 mg/kg | Part B: Sym004 12 mg/kg
Number analyzed (Participants) | 3 | 6 | 6 | 6 | 7
μg/mL/mg
  mAb992 | 0.306 (19.8) | 0.336 (23.5) | 0.346 (22.0) | 0.268 (19.1) | 0.284 (13.0)
  mAb1024 | 0.334 (8.4) | 0.353 (26.0) | 0.334 (13.4) | 0.317 (15.6) | 0.471 (58.7)

29. Secondary Outcome: Dose Nornamized Maximum Serum Concentration (Cmax) of Sym004 for the Weekly Regimen at Week 4: Multiple Dose
Description: Sym004 is a mixture of two mouse-human chimeric immunoglobulin G1 anti-epidermal growth factor receptor (EGFR) monoclonal antibodies (called monoclonal antibodies [mAb] 992 and mAb 1024). Here dose normalized Cmax are presented for both monoclonal antibodies. Dose normalized Cmax was calculated as Cmax/Dose. Weekly dosing cohorts (Part A: Sym004 6 mg/kg, Part A: Sym004 9/6 mg/kg, Part A: Sym004 12 mg/kg, Part B: Sym004 12 mg/kg) were only applicable for Week 4 assessment. Biweekly dosing cohort (Part A: Sym004 18 mg/kg) was not applicable for Week 4 assessment.
Time Frame: Pre-infusion, end of infusion, 4, 8, 12, 24 hours post-infusion at Week 4
Population: as for outcome 25
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL/mg
Arm/Group | Part A: Sym004 6 mg/kg | Part A: Sym004 9/6 mg/kg | Part A: Sym004 12 mg/kg | Part B: Sym004 12 mg/kg
Number analyzed (Participants) | 3 | 6 | 6 | 6
μg/mL/mg
  mAb992 | 0.486 (4.4) | 0.524 (31.4) | 0.516 (18.4) | 0.466 (12.8)
  mAb1024 | 0.570 (7.1) | 0.553 (32.3) | 0.629 (12.9) | 0.752 (24.3)

30. Secondary Outcome: Dose Normalized Maximum Serum Concentration (Cmax) of Sym004 for the Biweekly Regimen at Week 5: Multiple Dose
Description: Sym004 is a mixture of two mouse-human chimeric immunoglobulin G1 anti-epidermal growth factor receptor (EGFR) monoclonal antibodies (called monoclonal antibodies [mAb] 992 and mAb 1024). Here dose normalized Cmax are presented for both monoclonal antibodies. Weekly dosing cohorts (Part A: Sym004 6 mg/kg, Part A: Sym004 9/6 mg/kg, Part A: Sym004 12 mg/kg, Part B: Sym004 12 mg/kg) were not applicable for Week 5 assessment. Biweekly dosing cohort (Part A: Sym004 18 mg/kg) was only applicable for Week 5 assessment. Dose normalized Cmax was calculated as Cmax/Dose.
Time Frame: Pre-infusion, end of infusion, 4, 8, 12, 24 hours post-infusion at Week 5
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL/mg
Arm/Group | Part A: Sym004 18 mg/kg
Number analyzed (Participants) | 6
μg/mL/mg
  mAb992 | 0.318 (25.0)
  mAb1024 | 0.380 (20.2)

31. Secondary Outcome: Trough Concentrations (Ctrough) of Sym004
Description: Sym004 is a mixture of two mouse-human chimeric immunoglobulin G1 anti-epidermal growth factor receptor (EGFR) monoclonal antibodies (called monoclonal antibodies [mAb] 992 and mAb 1024). Ctrough are presented for both monoclonal antibodies.
Time Frame: Pre-infusion at Week 2, 3, 5, 6, 7, 8, End of Trial (up to 41.1 weeks) and Follow up (up to 45.1 Weeks)
Population: The PK Analysis Set consisted of all subjects (from Parts A and B) who received at least 1 administration of Sym004 and who provided sufficient data for a concentration time profile for Sym004. Here "Number of Participants Analyzed" =subjects who were evaluable for this outcome and "n" =subjects who were evaluable for specified time frame.
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Part A: Sym004 6 mg/kg | Part A: Sym004 9/6 mg/kg | Part A: Sym004 12 mg/kg | Part A: Sym004 18 mg/kg | Part B: Sym004 12 mg/kg
Number analyzed (Participants) | 3 | 6 | 6 | 6 | 29
μg/mL
  mAb992 Week 2 pre-dose (n= 3, 6, 6, 6, 29) | 8.38333 (2.562935) | 16.3617 (7.384964) | 29.4483 (9.716758) | 45.1117 (17.24716) | 20.1517 (8.411459)
  mAb992 Week 3 pre-dose (n= 3, 6, 5, 6, 26) | 19.8700 (9.570564) | 16.7033 (8.283479) | 57.7280 (29.34743) | 15.3600 (6.817337) | 32.6969 (12.62782)
  mAb992 Week 5 pre-dose (n= 2, 5, 6, 0, 23) | NA (NA) — Mean and standard deviation were not estimable if evaluable subjects were less than 3 as per the planned decision because only 2 collected values were not sufficient to calculate a reliable estimation | 22.9260 (11.37231) | 66.0267 (37.84088) | NA (NA) — No subjects were evaluable hence the parameter at specified time point was not analyzed. | 71.0739 (67.33365)
  mAb992 Week 6 pre-dose (n= 3, 5, 5, 4, 21) | 25.5833 (21.14422) | 26.3340 (13.43829) | 92.4920 (47.20264) | 64.3750 (20.56197) | 53.2224 (30.76489)
  mAb992 Week 7 pre-dose (n= 2, 4, 4, 4, 21) | NA (NA) — Mean and standard deviation were not estimable if evaluable subjects were less than 3 as per the planned decision because only 2 collected values were not sufficient to calculate a reliable estimation | 25.7500 (16.36742) | 70.9875 (61.05280) | 36.1700 (7.608184) | 66.1524 (65.22446)
  mAb992 Week 8 pre-dose (n= 2, 4, 3, 2, 12) | NA (NA) — Mean and standard deviation were not estimable if evaluable subjects were less than 3 as per the planned decision because only 2 collected values were not sufficient to calculate a reliable estimation | 24.8650 (13.70631) | 122.283 (79.73053) | NA (NA) — Mean and standard deviation were not estimable if evaluable subjects were less than 3 as per the planned decision because only 2 collected values were not sufficient to calculate a reliable estimation | 60.4542 (25.37663)
  mAb992 End of Trial(up to 41.1weeks)(n=3,6,6,6,27) | NA (NA) — Data could not be estimated as it was below lower limit of quantitation (LLOQ) for mAb992 (LLOQ: 0.5 μg/mL) | NA (NA) — Data could not be estimated as it was below lower limit of quantitation (LLOQ) for mAb992 (LLOQ: 0.5 μg/mL) | 13.8400 (32.25929) | 1.24833 (2.197339) | 5.63333 (11.64986)
  mAb992 Follow up (up to 45.1 Weeks)(n=1,2,3,4,19) | NA (NA) — Mean and standard deviation were not estimable if evaluable subjects were less than 3 as per the planned decision because only 2 collected values were not sufficient to calculate a reliable estimation | NA (NA) — Mean and standard deviation were not estimable if evaluable subjects were less than 3 as per the planned decision because only 2 collected values were not sufficient to calculate a reliable estimation | NA (NA) — Data could not be estimated as it was below lower limit of quantitation (LLOQ) for mAb992 (LLOQ: 0.5 μg/mL) | NA (NA) — Data could not be estimated as it was below lower limit of quantitation (LLOQ) for mAb992 (LLOQ: 0.5 μg/mL) | NA (NA) — Data could not be estimated as it was below lower limit of quantitation (LLOQ) for mAb992 (LLOQ: 0.5 μg/mL)
  mAb1024 Week 2 pre-dose (n= 3, 6, 6, 6, 29) | 10.6767 (2.688128) | 20.2433 (8.704451) | 38.7017 (12.01645) | 58.6967 (17.29509) | 27.8641 (12.33288)
  mAb1024 Week 3 pre-dose (n= 3, 6, 5, 6, 26) | 23.8000 (9.525382) | 22.7517 (14.69928) | 69.9460 (21.36079) | 24.7000 (11.16315) | 44.6531 (17.91820)
  mAb1024 Week 5 pre-dose (n= 2, 5, 6, 0, 23) | NA (NA) — Mean and standard deviation were not estimable if evaluable subjects were less than 3 as per the planned decision because only 2 collected values were not sufficient to calculate a reliable estimation | 31.8900 (17.43852) | 98.6550 (46.85021) | NA (NA) — No subjects were evaluable hence the parameter at specified time point was not analyzed. | 82.6235 (49.01981)
  mAb1024 Week 6 pre-dose (n= 3, 5, 5, 4, 21) | 31.8700 (23.97075) | 35.2440 (18.90163) | 128.858 (41.31495) | 90.9275 (26.82442) | 80.0024 (35.72029)
  mAb1024 Week 7 pre-dose (n= 2, 4, 4, 4, 21) | NA (NA) — Mean and standard deviation were not estimable if evaluable subjects were less than 3 as per the planned decision because only 2 collected values were not sufficient to calculate a reliable estimation | 36.1125 (24.42487) | 107.843 (76.48666) | 54.9275 (13.15679) | 94.4729 (52.58200)
  mAb1024 Week 8 pre-dose (n= 2, 4, 3, 2, 12) | NA (NA) — Mean and standard deviation were not estimable if evaluable subjects were less than 3 as per the planned decision because only 2 collected values were not sufficient to calculate a reliable estimation | 34.6050 (19.49550) | 166.207 (52.87010) | NA (NA) — Mean and standard deviation were not estimable if evaluable subjects were less than 3 as per the planned decision because only 2 collected values were not sufficient to calculate a reliable estimation | 93.0283 (47.35483)
  mAb1024End of Trial(up to 41.1weeks)(n=3,6,6,6,27) | NA (NA) — Data could not be estimated as it was below lower limit of quantitation (LLOQ) for mAb1024 (LLOQ: 0.5 μg/mL) | NA (NA) — Data could not be estimated as it was below lower limit of quantitation (LLOQ) for mAb1024 (LLOQ: 0.5 μg/mL) | 25.4667 (58.32014) | 3.73333 (6.795639) | 11.2478 (19.88056)
  mAb1024 Follow up (up to 45.1 Weeks)(n=1,2,3,4,19) | NA (NA) — Mean and standard deviation were not estimable if evaluable subjects were less than 3 as per the planned decision because only 2 collected values were not sufficient to calculate a reliable estimation | NA (NA) — Mean and standard deviation were not estimable if evaluable subjects were less than 3 as per the planned decision because only 2 collected values were not sufficient to calculate a reliable estimation | NA (NA) — Data could not be estimated as it was below lower limit of quantitation (LLOQ) for mAb1024 (LLOQ: 0.5 μg/mL) | NA (NA) — Data could not be estimated as it was below lower limit of quantitation (LLOQ) for mAb1024 (LLOQ: 0.5 μg/mL) | NA (NA) — Data could not be estimated as it was below lower limit of quantitation (LLOQ) for mAb1024 (LLOQ: 0.5 μg/mL)

32. Secondary Outcome: Time to Reach Maximum Concentration (Tmax) of Sym004 at Week 1: Single Dose
Description: Sym004 is a mixture of two mouse-human chimeric immunoglobulin G1 anti-epidermal growth factor receptor (EGFR) monoclonal antibodies (called monoclonal antibodies [mAb] 992 and mAb 1024). Tmax are presented for both monoclonal antibodies.
Time Frame: Pre-infusion, end of infusion, 4, 8, 12, 24, 48 hours post-infusion at Week 1
Population: as for outcome 25
Measure: Median (Full Range); unit: hours
Arm/Group | Part A: Sym004 6 mg/kg | Part A: Sym004 9/6 mg/kg | Part A: Sym004 12 mg/kg | Part A: Sym004 18 mg/kg | Part B: Sym004 12 mg/kg
Number analyzed (Participants) | 3 | 6 | 6 | 6 | 7
hours
  mAb992 | 2.07 [2.0 to 14] | 5.12 [3.1 to 7.2] | 5.73 [3.0 to 11.0] | 7.21 [3.2 to 15.0] | 6.30 [3.2 to 11.0]
  mAb1024 | 2.05 [2.0 to 2.1] | 7.20 [3.2 to 11] | 6.66 [3.1 to 11.0] | 7.15 [3.2 to 7.6] | 7.13 [3.2 to 11.0]

33. Secondary Outcome: Time to Reach Maximum Concentration (Tmax) of Sym004 for the Weekly Regimen at Week 4: Multiple Dose
Description: Sym004 is a mixture of two mouse-human chimeric immunoglobulin G1 anti-epidermal growth factor receptor (EGFR) monoclonal antibodies (called monoclonal antibodies [mAb] 992 and mAb 1024). Tmax are presented for both monoclonal antibodies. Weekly dosing cohorts (Part A: Sym004 6 mg/kg, Part A: Sym004 9/6 mg/kg, Part A: Sym004 12 mg/kg, Part B: Sym004 12 mg/kg) were only applicable for Week 4 assessment. Biweekly dosing cohort (Part A: Sym004 18 mg/kg) was not applicable for Week 4 assessment.
Time Frame: Pre-infusion, end of infusion, 4, 8, 12, 24 hours post-infusion at Week 4
Population: as for outcome 25
Measure: Median (Full Range); unit: hours
Arm/Group | Part A: Sym004 6 mg/kg | Part A: Sym004 9/6 mg/kg | Part A: Sym004 12 mg/kg | Part B: Sym004 12 mg/kg
Number analyzed (Participants) | 3 | 6 | 6 | 6
hours
  mAb992 | 10.1 [6.0 to 14] | 5.94 [2.325 to 9.0] | 9.13 [7.1 to 11.0] | 5.13 [2.9 to 11.0]
  mAb1024 | 2.07 [2.0 to 2.1] | 6.13 [2.0 to 18.0] | 5.18 [3.0 to 7.3] | 7.10 [3.1 to 11.0]

34. Secondary Outcome: Time to Reach Maximum Concentration (Tmax) of Sym004 for the Biweekly Regimen at Week 5: Multiple Dose
Description: Sym004 is a mixture of two mouse-human chimeric immunoglobulin G1 anti-epidermal growth factor receptor (EGFR) monoclonal antibodies (called monoclonal antibodies [mAb] 992 and mAb 1024). Tmax are presented for both monoclonal antibodies. Weekly dosing cohorts (Part A: Sym004 6 mg/kg, Part A: Sym004 9/6 mg/kg, Part A: Sym004 12 mg/kg, Part B: Sym004 12 mg/kg) were not applicable for Week 5 assessment. Biweekly dosing cohort (Part A: Sym004 18 mg/kg) was only applicable for Week 5 assessment.
Time Frame: Pre-infusion, end of infusion, 4, 8, 12, 24 hours post-infusion at Week 5
Population: as for outcome 7
Measure: Median (Full Range); unit: hours
Arm/Group | Part A: Sym004 18 mg/kg
Number analyzed (Participants) | 6
hours
  mAb992 | 7.03 [3.1 to 11.0]
  mAb1024 | 5.28 [3.1 to 11.0]

35. Secondary Outcome: Percentage of Subjects With Best Overall Response
Description: Percentage of subjects with best overall response (defined as confirmed CR or PR) according to Response Evaluation Criteria in Solid Tumors (RECIST Version 1.1) was reported. CR was defined as disappearance of all target and all non-target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 millimiter (mm). PR was defined as at least a 30% decrease in sum of diameters of target lesions, taking as reference the baseline sum diameters. Confirmed CR or PR was defined as the response that was confirmed at an interval of at least 4 weeks.
Time Frame: Week 7 and thereafter every 6 weeks, up to 4 weeks after last dose for Part A or up to 8 weeks after the last dose for Part B (up to 45.1 Weeks)
Population: Efficacy Analysis Set consisted of all subjects (from Parts A and B) who received at least 1 administration of Sym004 and who had baseline tumor assessment and at least 1 tumor assessment according to RECISTv1.1 after first dose of trial medication.
Measure: Number; unit: percentage of subjects
Arm/Group | Part A: Sym004 6 mg/kg | Part A: Sym004 9/6 mg/kg | Part A: Sym004 12 mg/kg | Part A: Sym004 18 mg/kg | Part B: Sym004 12 mg/kg
Number analyzed (Participants) | 3 | 6 | 6 | 6 | 30
percentage of subjects
  CR | 0 | 0 | 0 | 0 | 0
  PR | 0 | 0 | 33.3 | 0 | 16.7

36. Secondary Outcome: Duration of Overall Response
Description: The duration of overall response was measured from the time measurement criteria were first met for CR or PR (whichever was first recorded) until the first date that recurrent or progressive disease was objectively documented. CR was defined as disappearance of all target and all non-target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. PR was defined as at least a 30% decrease in sum of diameters of target lesions, taking as reference the baseline sum diameters. Confirmed CR or PR was defined as the response that was confirmed at an interval of at least 4 weeks.
Time Frame: Week 7 and thereafter every 6 weeks until the first date of objectively documented recurrent or progressive disease, up to 45.1 Weeks
Population: Efficacy Analysis Set consisted of all subjects (from Parts A and B) who received at least 1 administration of Sym004 and who had baseline tumor assessment and at least 1 tumor assessment according to RECISTv1.1 after first dose of trial medication. Here, "Number of Participants Analyzed" signifies those subjects who achieved confirmed CR or PR.
Measure: Median (Full Range); unit: Weeks
Arm/Group | Part A: Sym004 6 mg/kg | Part A: Sym004 9/6 mg/kg | Part A: Sym004 12 mg/kg | Part A: Sym004 18 mg/kg | Part B: Sym004 12 mg/kg
Number analyzed (Participants) | 0 | 0 | 2 | 0 | 5
Weeks |  |  | 25.85 [24.6 to 27.1] |  | 10.40 [8.1 to 22.1]

37. Secondary Outcome: Percentage of Subjects With Disease Control
Description: Percentage of subjects with disease control (defined as confirmed CR, confirmed PR, or confirmed SD) ) according to RECIST Version 1.1 was reported. CR: disappearance of all target and all non-target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. PR: at least a 30% decrease in sum of diameters of target lesions, taking as reference the baseline sum diameters. PD: at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study) or unequivocal progression of existing non-target lesions. SD: neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study. Confirmed CR or PR: response confirmed at an interval of at least 4 weeks. Confirmed SD: response confirmed at an interval of at least 6 weeks.
Time Frame: as for outcome 35
Population: as for outcome 35
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Part A: Sym004 6 mg/kg | Part A: Sym004 9/6 mg/kg | Part A: Sym004 12 mg/kg | Part A: Sym004 18 mg/kg | Part B: Sym004 12 mg/kg
Number analyzed (Participants) | 3 | 6 | 6 | 6 | 30
percentage of subjects | 66.7 [9.4 to 99.2] | 66.7 [22.3 to 95.7] | 50.0 [11.8 to 88.2] | 16.7 [0.4 to 64.1] | 56.7 [37.4 to 74.5]

38. Secondary Outcome: Duration of Disease Control
Description: Duration of disease control measured from the time measurement criteria were first met for CR, PR, or SD (whichever was first recorded) until the first date that recurrent or progressive disease was objectively documented. CR: disappearance of all target and all non-target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. PR: at least a 30% decrease in sum of diameters of target lesions, taking as reference the baseline sum diameters. PD: at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study) or unequivocal progression of existing non-target lesions. SD: neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study.
Time Frame: as for outcome 36
Population: Efficacy Analysis Set consisted of all subjects (from Parts A and B) who received at least 1 administration of Sym004 and who had baseline tumor assessment and at least 1 tumor assessment according to RECISTv1.1 after first dose of trial medication. Here, "Number of Participants Analyzed" signifies those subjects who achieved disease control.
Measure: Median (Full Range); unit: Weeks
Arm/Group | Part A: Sym004 6 mg/kg | Part A: Sym004 9/6 mg/kg | Part A: Sym004 12 mg/kg | Part A: Sym004 18 mg/kg | Part B: Sym004 12 mg/kg
Number analyzed (Participants) | 2 | 4 | 3 | 1 | 17
Weeks | 6.10 [6.1 to 6.1] | 5.35 [4.0 to 6.1] | 24.60 [4.1 to 27.1] | 6.10 [6.1 to 6.1] | 5.90 [0.1 to 22.1]

39. Secondary Outcome: Time to Progression
Description: Time to progression was defined as the time from date of subject enrollment until the date that disease progression was objectively documented. TTP estimated using the Kaplan-Meier estimates. TTP was planned to be reported for Part B alone and Part A/B combined reporting arms.
Time Frame: Time from enrollment until the date of objectively documented disease progression or death, up to 45.1 Weeks
Population: as for outcome 35
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Part A and B Combined: All subjects who were included in Part A and Part B. Sym004 administered by intravenous infusion at a dose of 6 mg/kg weekly, or 9 mg/kg at Week 1 followed by a maintenance dose of 6 mg/kg weekly, or 12 mg/kg weekly, or 18 mg/kg biweekly in Part A or 12 mg/kg by intravenous infusion weekly in Part B until unacceptable toxicity, disease progression, or consent withdrawal, or until the subject met any of the criteria for treatment or trial discontinuation.
Arm/Group | Part B: Sym004 12 mg/kg | Part A and B Combined
Number analyzed (Participants) | 30 | 51
months | 2.37 [1.38 to 3.68] | 2.33 [1.41 to 2.79]

40. Secondary Outcome: Progression-free Survival Time
Description: The Progression-free survival time was measured from the date of subject enrollment until the date that disease progression was objectively documented or death. Progression-free survival time estimated with using the Kaplan-Meier method. Progression-free survival time was planned to be reported for Part B alone and Part A/B combined reporting arms.
Time Frame: Time from enrollment until the date of objectively documented disease progression or death, up to 45.1 Weeks
Population: as for outcome 35
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Part B: Sym004 12 mg/kg | Part A and B Combined
Number analyzed (Participants) | 30 | 51
months | 2.12 [1.38 to 2.83] | 2.30 [1.41 to 2.79]

41. Secondary Outcome: Anti-drug Antibody Titers
Time Frame: Week 1 (pre-dose) up to Follow-up assessment (up to maximum 45.1 Weeks)
Population: Anti-drug Antibody (ADA) titer could not be estimated because there were no subjects who were confirmed to have ADA positive test results during the confirmatory analysis.
Arm/Group | Part A: Sym004 6 mg/kg | Part A: Sym004 9/6 mg/kg | Part A: Sym004 12 mg/kg | Part A: Sym004 18 mg/kg | Part B: Sym004 12 mg/kg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

42. Secondary Outcome: Percentage of Participants With Epidermal Growth Factor Receptor (EGFR) Expression in Skin Tissues by Immunohistochemistry (IHC)
Description: IHC is a staining process performed on fresh/frozen cancer tissue. IHC is used to show whether or not the cancer cells have Human Epidermal Growth Receptor (HER2) and/or hormone receptors on their surface. A value designated the IHC score was derived by summing the percentages of cells staining at each intensity multiplied by the weighted intensity of staining (0, 1+, 2+, 3+: 3+ indicates the strongest staining, 2+ indicates medium staining, 1+ indicates weak staining, and 0 indicates no staining). Minimum score of 0 to a maximum score of 300; the maximum score indicates the strongest expression.
Time Frame: Week 1 (pre-dose), Week 4 and Week 5
Population: The Biomarker analysis set consisted of all subjects who received at least 1 administration of Sym004 and who had at least 1 biomarker evaluation.
Measure: Number; unit: percentage of subjects
Arm/Group | Part A: Sym004 6 mg/kg | Part A: Sym004 9/6 mg/kg | Part A: Sym004 12 mg/kg | Part A: Sym004 18 mg/kg | Part B: Sym004 12 mg/kg
Number analyzed (Participants) | 3 | 6 | 6 | 6 | 13
percentage of subjects
  Week 1: 0 Score | 0.0 | 0.0 | 0.0 | 0.0 | 7.7
  Week 1: greater than (>) 0-less than(<) 100 Score | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Week 1: 100 - <200 Score | 33.3 | 0.0 | 16.7 | 0.0 | 0.0
  Week 1: 200 - 300 Score | 66.7 | 83.3 | 83.3 | 100.0 | 76.9
  Week 1: Missing | 0.0 | 16.7 | 0.0 | 0.0 | 15.4
  Week 4: 0 Score | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Week 4: >0 - <100 Score | 0.0 | 0.0 | 0.0 | 0.0 | 15.4
  Week 4: 100 - <200 Score | 33.3 | 83.3 | 33.3 | 0.0 | 46.2
  Week 4: 200 - 300 Score | 66.7 | 16.7 | 66.7 | 0.0 | 23.1
  Week 4: Missing | 0.0 | 0.0 | 0.0 | 100.0 | 15.4
  Week 5: 0 Score | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Week 5: >0 - <100 Score | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Week 5: 100 - <200 Score | 0.0 | 0.0 | 0.0 | 16.7 | 0.0
  Week 5: 200 - 300 Score | 0.0 | 0.0 | 0.0 | 66.7 | 0.0
  Week 5: Missing | 100.0 | 100.0 | 100.0 | 16.7 | 100.0

43. Secondary Outcome: Percentage of Participants With EGFR Amplification Using Fluorescent in Situ Hybridization (FISH) Method.
Time Frame: Week 1 (pre-dose) and Week 4.
Population: as for outcome 42
Measure: Number; unit: percentage of subjects
Arm/Group | Part A: Sym004 6 mg/kg | Part A: Sym004 9/6 mg/kg | Part A: Sym004 12 mg/kg | Part A: Sym004 18 mg/kg | Part B: Sym004 12 mg/kg
Number analyzed (Participants) | 3 | 6 | 6 | 6 | 13
percentage of subjects
  Week 1: EGFR-FISH Positive | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Week 1: EGFR-FISH Negative | 0.0 | 0.0 | 0.0 | 0.0 | 53.8
  Week 1: missing | 100.0 | 100.0 | 100.0 | 100.0 | 46.2
  Week 4: EGFR-FISH Positive | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Week 4: EGFR-FISH Negative | 0.0 | 0.0 | 0.0 | 0.0 | 23.1
  Week 4: missing | 100.0 | 100.0 | 100.0 | 100.0 | 76.9

ADVERSE EVENTS:
Time Frame: Baseline up to 4 weeks after the last Sym004 administration, up to a maximum of 41.1 weeks
Arm/Group | Part A: Sym004 6 mg/kg | Part A: Sym004 9/6 mg/kg | Part A: Sym004 12 mg/kg | Part A: Sym004 18 mg/kg | Part B: Sym004 12 mg/kg
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/6 | 2/6 | 0/6 | 9/30
Other Adverse Events (participants affected / at risk) | 3/3 | 6/6 | 6/6 | 6/6 | 30/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: Sym004 6 mg/kg (N=3) | Part A: Sym004 9/6 mg/kg (N=6) | Part A: Sym004 12 mg/kg (N=6) | Part A: Sym004 18 mg/kg (N=6) | Part B: Sym004 12 mg/kg (N=30)
Cardiac arrest (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Lung infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Dyspnoea at rest (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Pulmonary fistula (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Venous thrombosis limb (Vascular disorders) | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: Sym004 6 mg/kg (N=3) | Part A: Sym004 9/6 mg/kg (N=6) | Part A: Sym004 12 mg/kg (N=6) | Part A: Sym004 18 mg/kg (N=6) | Part B: Sym004 12 mg/kg (N=30)
Anaemia (Blood and lymphatic system disorders) | 2 | 0 | 1 | 0 | 1
Eosinophilia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 1
Lymphopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 2
Palpitations (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Conjunctival hyperaemia (Eye disorders) | 0 | 0 | 1 | 0 | 0
Eye discharge (Eye disorders) | 0 | 0 | 0 | 0 | 2
Cheilitis (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 7
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 3 | 1 | 4
Gingival bleeding (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 3
Stomatitis (Gastrointestinal disorders) | 1 | 3 | 2 | 0 | 10
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 1
Face oedema (General disorders) | 0 | 1 | 1 | 0 | 3
Fatigue (General disorders) | 1 | 0 | 2 | 1 | 13
Malaise (General disorders) | 1 | 0 | 0 | 0 | 1
Oedema peripheral (General disorders) | 0 | 1 | 2 | 1 | 4
Pyrexia (General disorders) | 0 | 0 | 2 | 1 | 2
Conjunctivitis (Infections and infestations) | 0 | 1 | 1 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Lung infection (Infections and infestations) | 0 | 0 | 0 | 0 | 2
Paronychia (Infections and infestations) | 1 | 1 | 2 | 2 | 10
Peritonitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 2 | 2 | 2 | 9
Overdose (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1 | 2 | 1 | 5
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 1 | 1 | 5
Blood alkaline phosphatase increased (Investigations) | 1 | 1 | 0 | 0 | 3
Blood bilirubin increased (Investigations) | 1 | 0 | 1 | 1 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 1 | 0 | 1
Blood magnesium decreased (Investigations) | 0 | 0 | 0 | 0 | 2
Blood urine present (Investigations) | 0 | 0 | 0 | 0 | 3
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 0 | 0 | 4
Lymphocyte count decreased (Investigations) | 0 | 0 | 2 | 0 | 1
Platelet count decreased (Investigations) | 0 | 0 | 0 | 1 | 0
Weight decreased (Investigations) | 3 | 1 | 0 | 0 | 9
Weight increased (Investigations) | 0 | 0 | 2 | 1 | 3
White blood cell count decreased (Investigations) | 1 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 2 | 0 | 8
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 1
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 2
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1 | 3 | 2 | 8
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 6
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 2 | 0 | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 3 | 6 | 5 | 5 | 20
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 2
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 1 | 1 | 7
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 2
Peripheral motor neuropathy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 1 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 3
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 3
Proteinuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 3
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 3 | 6 | 6 | 5 | 23
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 2 | 0 | 4 | 17
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Hirsutism (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 2
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 5
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 11
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1 | 2 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 4
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 6
Skin atrophy (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 1
Skin fissures (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 0 | 1
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Flushing (Vascular disorders) | 0 | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No